CLINICAL TRIAL: NCT05100719
Title: The Role of Irritable Bowel Syndrome in Lactose Intolerance (LION Trial): Protocol of a Multicentre Randomized Controlled Clinical Trial
Brief Title: The Role of Irritable Bowel Syndrome in Lactose Intolerance (LION)
Acronym: LION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, József Czimmer, Divison of Gastroenterology, First Department of Medicine, Medical School, University of Pécs, Pécs, Hungary, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IV/4455-3/2021/EKU
Record Dates: First submitted 2021-09-29; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Irritable Bowel Syndrome; Lactose Intolerance; Lactose Malabsorption
Keywords: irritable bowel syndrome; lactose intolerance; lactose malabsorption; lactase; simethicone; alverine-citrate; placebo
MeSH Terms: conditions — Irritable Bowel Syndrome; Lactose Intolerance | interventions — mebeverine; Simethicone; Lactase

STUDY DESIGN:
Intervention Model Description: LION is a two-armed, randomized, double-blind, placebo-controlled, two-phase clinical trial. In the first phase, we will enroll 100 patients, the allocation ratio will be 1:1 (50 patinets in each arm). Then, an interim analysis will be performed to determine the appropriate sample size. During the interim analysis, if there is already significant difference (p<0.0294) between the arms, the recruitment will be considered completed; otherwise, recruitment will continue until the desired sample size is reached. If there is no hope for ascertaining significance, the study will be stopped.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alverine-citrate + simethicone and lactase (Active Comparator): Patients diagnosed with irritable bowel syndrome based on the ROME IV criteria will go through a lactase intolerance test (LTT) and (lactose H2 breath test) LHBT. Those who have positive LTT and LHBT will receive alverine-citrate + simethicone and lactase.
  Interventions: Drug: alverine-citrate + simethicone and lactase
- alverin-citrate + simethicone with placebo (Placebo Comparator): Patients diagnosed with irritable bowel syndrome based on the ROME IV criteria will go through a lactase intolerance test (LTT) and (lactose H2 breath test) LHBT. Those who have positive LTT and LHBT will receive alverine-citrate + simethicone with placebo.
  Interventions: Drug: alverin-citrate + simethicone with placebo

INTERVENTIONS:
Drug: alverine-citrate + simethicone and lactase — Patients who randomized in the first arm are treated with alverine-citrate + simethicone and lactase.
  Other Names: lactase
  Arms: alverine-citrate + simethicone and lactase
Drug: alverin-citrate + simethicone with placebo — Patients in the second arm receive alverin-citrate + simethicone with placebo without lactase.
  Other Names: placebo
  Arms: alverin-citrate + simethicone with placebo

SUMMARY:
Irritable bowel syndrome (IBS) is a functional gastrointestinal disease. There is no well-defined pharmacological treatment. This clinical trial is a prospective, double-blind, two-armed randomized controlled, single-center trial. It is created to examine the role of IBS in patients with lactose intolerance. IBS patients undergo lactose H2 breath test (LHBT) and lactose tolerance test (LTT). Those with positive LTT and LHBT will be randomized into two groups: alverine-citrate + simethicone and lactase group (1) or alverin-citrate + simethicone with the placebo group (2). The goal of this study is to compare the lactase enzyme with placebo in IBS patients with lactose intolerance.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is one of the most frequently diagnosed gastroenterological disorders and can lead to significant deterioration of quality of life and an increase in health care and societal costs. Patients with lactose intolerance are unable to fully digest lactose caused by lactose malabsorption. The undigested lactose moves into the large intestine, fermented by bacteria, and causes bloating, gas, and diarrhea symptoms. The two, most frequently used diagnostic methods are the lactose H2 breath test (LHBT) and the lactose tolerance test (LTT). The restriction of lactose input or the replacement of the lactase enzyme can lead to the relief of the symptoms. Lactose intolerance is a common disorder among patients with IBS, it is more frequent than in the general population.

There are no studies that assess the link between lactose intolerance and IBS. Our primary objective is the examination of the relationship between lactose intolerance and IBS with or without the replacement of lactase enzyme. Our secondary objectives are to compare the lactase/beta-galactosidase enzyme replacement with placebo with the evaluation of a TSS (Total symptom score), VAS (Visual Analog Scale), QoL (Quality of life) questionnaires. The other secondary outcomes are to compare the severity of baseline symptoms during and after lactose administration.

Patients diagnosed with IBS according to the Rome IV criteria will test with LTT and LHBT.

Who has positive LTT and LHBT will randomize into two groups: (1) alverine-citrate + simethicone and lactase; (2) alverin-citrate + simethicone with placebo.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* patients diagnosed with irritable bowel syndrome based on the ROME IV. criteria
* positive LHBT (lactose H2 breath test) and LTT (lactose tolerance test) results
* negative abdominal ultrasound/CAT scan/MRI results within one year
* signed the informed consent

Exclusion Criteria:

* organic gastroenterological disorders which can explain symptoms (e.g. positive serological screening: anti-gliadin IgG / IgA, anti-tissue transglutaminase IgG / IgA, high level of fecal calprotectin tested by endoscopy or positive colonoscopy for IBD, currently active diverticulitis
* Alarm symptoms: fever (> 38 Co), anaemia (Hgb < 120 g/l), unintended weight loss (> 4.5 kg / 3 months), gastrointestinal bleeding (hematemesis, hematochesia, melena)
* cardiac failure (NYHA III-IV)
* liver cirrhosis (Child-Pugh C)
* active malignancy
* major abdominal surgery in the history
* pregnant or breastfeeding women
* any circumstances which can lead to false results of LHBT and LTT: cigarette smoking or physical exercise within 2 hours before the test, ingestion of dietary fibers on the evening before the test, recent use of antibiotics, lung disease, baseline H2 concentration in the exhaled air is higher than 20 ppm, not properly treated diabetes mellitus, following lactose restricted or another special diet within 1 week prior to study enrolment (ingestion of less than 12 g lactose - less than 250 ml milk - per day)
* small intestinal bacterial overgrowth (SIBO): if there is a rapid increase of H2 level in the exhaled air (≥20 ppm above baseline within 90 minutes), SIBO is suspected and antibiotic therapy will be started (peroral rifaximin for 5 days) after negative Helicobacter pylori serology. After this procedure, lactulose H2 breath test will be performed to exclude SIBO (≥20 ppm H2 rise only after 90 min). In case of negative lactulose H2 breath test, another LHBT will be carried out
* slow oro-cecal transit: clinical signs and typical findings on the tests (the LHBT is normal, but the increase of blood glucose level is less than 1.1 mmol/l and/or no H2 rise during lactulose H2 breath test)
* milk allergy (positive IgE test)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
change of the symptoms measured by TSS (total symptom score) | The one- and two-week total symptom score (TSS) change compared to baseline value.
  The primary outcome is the number of enrolled patients with significant improvement in each treatment arm. Significant improvement is considered if there is >50% reduction in the TSS, compared to the baseline symptoms.

SECONDARY OUTCOMES:
improvement in stool consistency | The two time points at which the measurement is assessed are the time of enrollment and after 2 weeks.
  stool consistency score of <5, according to the Bristol stool chart
the absence of a bowel movement | The three time points at which the measurement is assessed are the time of enrollment, after 1 and 2 weeks.
  The absence of a bowel movement is accompanied by an improvement of ≥30 mm in the VAS (visual analogue scale) for the worst abdominal pain.
relief of IBS-related bloating | The three time points at which the measurement is assessed are the time of enrollment, after 1 and 2 weeks.
  The number of patients with acceptable relief of IBS-related bloating determined by a questionnaire, from the response (yes or no) compare to the baseline IBS-related bloating.
Onset and duration of relief of bloating | The three time points at which the measurement is assessed are the time of enrollment, after 1 and 2 weeks.
  Onset and duration of relief of bloating is measured by a questionnaire.
incidence of Small intestinal bacterial overgrowth (SIBO) | At the time of patient enrollment and after two weeks of treatments this test will be carried out again.
  Early (within 90 minutes), significant (≥20 ppm) H2 rise during LHBT or lactulose breath test compared to the baseline value.
results of LHBT and LTT | At the time of patient enrollment and after two weeks of treatments LHBT and LTT will be carried out again.
  Results of LHBT (lactose H2 breath test) and LTT (lactose tolerance test).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Translational Medicine, University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately following publication. No end date
Access Criteria: With anyone who wishes to access the data. For any purpose of analyses.

REFERENCES:
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Borghini R, Donato G, Alvaro D, Picarelli A. New insights in IBS-like disorders: Pandora's box has been opened; a review. Gastroenterol Hepatol Bed Bench. 2017 Spring;10(2):79-89. PMID 28702130
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Muller-Lissner SA, Bollani S, Brummer RJ, Coremans G, Dapoigny M, Marshall JK, Muris JW, Oberndorff-Klein Wolthuis A, Pace F, Rodrigo L, Stockbrugger R, Vatn MH. Epidemiological aspects of irritable bowel syndrome in Europe and North America. Digestion. 2001;64(3):200-4. doi: 10.1159/000048862. PMID 11786669
- [Background] Drossman DA, Morris CB, Schneck S, Hu YJ, Norton NJ, Norton WF, Weinland SR, Dalton C, Leserman J, Bangdiwala SI. International survey of patients with IBS: symptom features and their severity, health status, treatments, and risk taking to achieve clinical benefit. J Clin Gastroenterol. 2009 Jul;43(6):541-50. doi: 10.1097/MCG.0b013e318189a7f9. PMID 19384249
- [Background] Agarwal N, Spiegel BM. The effect of irritable bowel syndrome on health-related quality of life and health care expenditures. Gastroenterol Clin North Am. 2011 Mar;40(1):11-9. doi: 10.1016/j.gtc.2010.12.013. PMID 21333898
- [Background] Dean BB, Aguilar D, Barghout V, Kahler KH, Frech F, Groves D, Ofman JJ. Impairment in work productivity and health-related quality of life in patients with IBS. Am J Manag Care. 2005 Apr;11(1 Suppl):S17-26. PMID 15926760
- [Background] Simren M, Svedlund J, Posserud I, Bjornsson ES, Abrahamsson H. Health-related quality of life in patients attending a gastroenterology outpatient clinic: functional disorders versus organic diseases. Clin Gastroenterol Hepatol. 2006 Feb;4(2):187-95. doi: 10.1016/s1542-3565(05)00981-x. PMID 16469679
- [Background] Bohn L, Storsrud S, Liljebo T, Collin L, Lindfors P, Tornblom H, Simren M. Diet low in FODMAPs reduces symptoms of irritable bowel syndrome as well as traditional dietary advice: a randomized controlled trial. Gastroenterology. 2015 Nov;149(6):1399-1407.e2. doi: 10.1053/j.gastro.2015.07.054. Epub 2015 Aug 5. PMID 26255043
- [Background] Hillila MT, Farkkila NJ, Farkkila MA. Societal costs for irritable bowel syndrome--a population based study. Scand J Gastroenterol. 2010 May;45(5):582-91. doi: 10.3109/00365521003637211. PMID 20166844
- [Background] Simren M, Barbara G, Flint HJ, Spiegel BM, Spiller RC, Vanner S, Verdu EF, Whorwell PJ, Zoetendal EG; Rome Foundation Committee. Intestinal microbiota in functional bowel disorders: a Rome foundation report. Gut. 2013 Jan;62(1):159-76. doi: 10.1136/gutjnl-2012-302167. Epub 2012 Jun 22. PMID 22730468
- [Background] Miller V, Hopkins L, Whorwell PJ. Suicidal ideation in patients with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2004 Dec;2(12):1064-8. doi: 10.1016/s1542-3565(04)00545-2. PMID 15625650
- [Background] Yang J, Fox M, Cong Y, Chu H, Zheng X, Long Y, Fried M, Dai N. Lactose intolerance in irritable bowel syndrome patients with diarrhoea: the roles of anxiety, activation of the innate mucosal immune system and visceral sensitivity. Aliment Pharmacol Ther. 2014 Feb;39(3):302-11. doi: 10.1111/apt.12582. Epub 2013 Dec 5. PMID 24308871
- [Background] Lomer MC, Parkes GC, Sanderson JD. Review article: lactose intolerance in clinical practice--myths and realities. Aliment Pharmacol Ther. 2008 Jan 15;27(2):93-103. doi: 10.1111/j.1365-2036.2007.03557.x. Epub 2007 Oct 23. PMID 17956597
- [Background] Suchy FJ, Brannon PM, Carpenter TO, Fernandez JR, Gilsanz V, Gould JB, Hall K, Hui SL, Lupton J, Mennella J, Miller NJ, Osganian SK, Sellmeyer DE, Wolf MA. National Institutes of Health Consensus Development Conference: lactose intolerance and health. Ann Intern Med. 2010 Jun 15;152(12):792-6. doi: 10.7326/0003-4819-152-12-201006150-00248. Epub 2010 Apr 19. No abstract available. PMID 20404261
- [Background] Misselwitz B, Pohl D, Fruhauf H, Fried M, Vavricka SR, Fox M. Lactose malabsorption and intolerance: pathogenesis, diagnosis and treatment. United European Gastroenterol J. 2013 Jun;1(3):151-9. doi: 10.1177/2050640613484463. PMID 24917953
- [Background] Monsbakken KW, Vandvik PO, Farup PG. Perceived food intolerance in subjects with irritable bowel syndrome-- etiology, prevalence and consequences. Eur J Clin Nutr. 2006 May;60(5):667-72. doi: 10.1038/sj.ejcn.1602367. PMID 16391571
- [Background] Di Stefano M, Miceli E, Mazzocchi S, Tana P, Moroni F, Corazza GR. Visceral hypersensitivity and intolerance symptoms in lactose malabsorption. Neurogastroenterol Motil. 2007 Nov;19(11):887-95. doi: 10.1111/j.1365-2982.2007.00973.x. Epub 2007 Aug 17. PMID 17973635
- [Background] Zhu Y, Zheng X, Cong Y, Chu H, Fried M, Dai N, Fox M. Bloating and distention in irritable bowel syndrome: the role of gas production and visceral sensation after lactose ingestion in a population with lactase deficiency. Am J Gastroenterol. 2013 Sep;108(9):1516-25. doi: 10.1038/ajg.2013.198. Epub 2013 Aug 6. PMID 23917444
- [Background] Vesa TH, Seppo LM, Marteau PR, Sahi T, Korpela R. Role of irritable bowel syndrome in subjective lactose intolerance. Am J Clin Nutr. 1998 Apr;67(4):710-5. doi: 10.1093/ajcn/67.4.710. PMID 9537618
- [Background] Vernia P, Di Camillo M, Marinaro V. Lactose malabsorption, irritable bowel syndrome and self-reported milk intolerance. Dig Liver Dis. 2001 Apr;33(3):234-9. doi: 10.1016/s1590-8658(01)80713-1. PMID 11407668
- [Background] Varju P, Gede N, Szakacs Z, Hegyi P, Cazacu IM, Pecsi D, Fabian A, Szepes Z, Vincze A, Tenk J, Balasko M, Rumbus Z, Garami A, Csupor D, Czimmer J. Lactose intolerance but not lactose maldigestion is more frequent in patients with irritable bowel syndrome than in healthy controls: A meta-analysis. Neurogastroenterol Motil. 2019 May;31(5):e13527. doi: 10.1111/nmo.13527. Epub 2018 Dec 17. PMID 30560578
- [Background] Yang J, Deng Y, Chu H, Cong Y, Zhao J, Pohl D, Misselwitz B, Fried M, Dai N, Fox M. Prevalence and presentation of lactose intolerance and effects on dairy product intake in healthy subjects and patients with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2013 Mar;11(3):262-268.e1. doi: 10.1016/j.cgh.2012.11.034. Epub 2012 Dec 13. PMID 23246646
- [Background] Bohmer CJ, Tuynman HA. The clinical relevance of lactose malabsorption in irritable bowel syndrome. Eur J Gastroenterol Hepatol. 1996 Oct;8(10):1013-6. doi: 10.1097/00042737-199610000-00015. PMID 8930569
- [Background] Vernia P, Ricciardi MR, Frandina C, Bilotta T, Frieri G. Lactose malabsorption and irritable bowel syndrome. Effect of a long-term lactose-free diet. Ital J Gastroenterol. 1995 Apr;27(3):117-21. PMID 7548919
- [Background] Lisker R, Solomons NW, Perez Briceno R, Ramirez Mata M. Lactase and placebo in the management of the irritable bowel syndrome: a double-blind, cross-over study. Am J Gastroenterol. 1989 Jul;84(7):756-62. PMID 2500848
- [Background] Hillila M, Farkkila MA, Sipponen T, Rajala J, Koskenpato J. Does oral alpha-galactosidase relieve irritable bowel symptoms? Scand J Gastroenterol. 2016 Jan;51(1):16-21. doi: 10.3109/00365521.2015.1063156. Epub 2015 Jul 2. PMID 26133538
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Hayase M, Hashitani H, Suzuki H, Kohri K, Brading AF. Evolving mechanisms of action of alverine citrate on phasic smooth muscles. Br J Pharmacol. 2007 Dec;152(8):1228-38. doi: 10.1038/sj.bjp.0707496. Epub 2007 Oct 15. PMID 17934514
- [Background] Ducrotte P, Grimaud JC, Dapoigny M, Personnic S, O'Mahony V, Andro-Delestrain MC. On-demand treatment with alverine citrate/simeticone compared with standard treatments for irritable bowel syndrome: results of a randomised pragmatic study. Int J Clin Pract. 2014 Feb;68(2):245-54. doi: 10.1111/ijcp.12333. Epub 2013 Oct 21. PMID 24147869
- [Result] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- See also: LION is designed and coordinated by the Centre for Translational Medicine (Medical School, University of Pécs). This link redirects to the official website of the institute. — http://tm-centre.org/